CLINICAL TRIAL: NCT05777161
Title: A Randomized-controlled Trial of Therapy for Children and Adolescents With Anxiety Disorders and Obsessive Compulsive Disorder (OCD)
Brief Title: A Trial of Parent-coached Exposure Therapy for Children With Anxiety Disorders and OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen Whiteside, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-008982
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Anxiety Disorders; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Anxiety Disorders; Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blind to condition. The integrity of the blind was evaluated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parent Coached Exposure Therapy-Individual (PCET-I) Group (Experimental): Subjects will receive six to 14 weekly sessions of individual Parent Coached Exposure Therapy
  Interventions: Behavioral: Parent Coached Exposure Therapy - Individualized
- Traditional Cognitive Behavior Therapy (CBT) Group (Active Comparator): Subjects will receive 6 to 14 weekly sessions of individual Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavior Therapy
- Parent Coached Exposure Therapy-5day Intensive (PCET-5day) Group (removed from study) (Experimental): Subjects will receive 5 day (nine sessions) of group-based Parent Coached Exposure Therapy delivered within a span of five days (Monday through Friday), followed by 5 weeks of self-care
  Interventions: Behavioral: Parent Coached Exposure Therapy - Group (removed from study)

INTERVENTIONS:
Behavioral: Parent Coached Exposure Therapy - Individualized — Subject and parent begin by working with a therapist to create an individualized fear hierarchy consisting of situations and stimuli that produce anxiety for the child, gradually progressing from less anxiety to more anxiety.
  Other Names: PCET-I
  Arms: Parent Coached Exposure Therapy-Individual (PCET-I) Group
Behavioral: Cognitive Behavior Therapy — Subjects will work with a therapist using anxiety management strategies to address thoughts, feelings, and behaviors.
  Other Names: CBT
  Arms: Traditional Cognitive Behavior Therapy (CBT) Group
Behavioral: Parent Coached Exposure Therapy - Group (removed from study) — Subjects and parents will work in a group setting to receive exposure therapy consisting of situations and stimuli that produce anxiety for the child, gradually progressing from less anxiety to more anxiety.
  Other Names: PCET
  Arms: Parent Coached Exposure Therapy-5day Intensive (PCET-5day) Group (removed from study)

SUMMARY:
The purpose of this study is to examine the effectiveness of parent coached exposure therapy (PCET) and standard cognitive behavioral therapy (CBT) in treating childhood anxiety disorders and obsessive compulsive disorder (OCD).

DETAILED DESCRIPTION:
The purpose of this study is to examine the effectiveness of parent coached exposure therapy (PCET) through baseline comparisons, to compare effectiveness of individual PCET and individual standard cognitive behavioral therapy (CBT), to compare efficiency of individual PCET and individual standard CBT, to compare effectiveness of group intensive PCET, individual PCET, and individual standard CBT, and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Have a DSM-5 anxiety disorder diagnosis, including generalized anxiety disorder, obsessive compulsive disorder, panic disorder, agoraphobia, separation anxiety disorder, social and specific phobias, as assessed on the relevant modules of the (MINI-Kids; (Sheehan et al., 2010) by study staff in the PADC.
* Be appropriate for the PADC standard outpatient therapy program, and be interested in starting outpatient therapy,
* Have the anxiety disorder as their primary diagnosis,
* If taking a selective serotonin reuptake inhibitor, SNRI, tricyclic, or antipsychotic medication, had no medication changes made at least 8 weeks prior to initiating participation in the study and agree to no changes during the 12 weeks of the study.

Exclusion Criteria:

* History of and/or current psychosis, autism, bipolar disorder, or current suicidality, or eating disorder as assessed during the initial clinical interview and all available clinical information.
* Current positive diagnosis in the child's caregiver of mental retardation, psychosis, or other psychiatric disorders or conditions that would limit his/her ability to understand CBT and follow-through with treatment directives (based on clinical interview).
* Secondary diagnosis of oppositional defiant disorder or major depression of sufficient severity to prevent anxiety treatment.
* Severity of symptoms that warrant higher level of care (i.e. intensive, residential, IOP, inpatient)
* Family is unable to attend weekly sessions (i.e. geographical or scheduling barriers)
* History of good quality exposure or CBT.

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in symptom severity per blinded independent evaluator | Baseline, mid-treatment (after 6 sessions), post-treatment (approximately 14 weeks)
  Measured by the Clinical Global Impression Scale (GCI-S) rating of severity of psychopathology ranging from 1 (not at all ill) to 7 (extremely ill), with a score of 1 or 2 reflecting no to minimal symptoms
Treatment efficiency | post-treatment (approximately 14 weeks)
  Number of appointments attended

SECONDARY OUTCOMES:
Change in anxiety symptoms per blinded independent evaluator | Baseline, mid-treatment (after 6 sessions), post-treatment (approximately 14 weeks)
  Pediatric Anxiety Rating Scale consisting of 5 items rated from 0 (no symptoms) to 5 (most severe) summed for a total score ranging from 0 (no symptoms) to 25 (most severe).
Change in symptom severity per parent | Baseline, mid-treatment (after 6 sessions), post-treatment (approximately 14 weeks)
  Spence Children's Anxiety Scale parent-report consisting of 38 items rated from 0 (never) to 3 (always) summed to a total score of 0 (no symptoms) to 108 (most severe).
Change in symptom severity per child | Baseline, mid-treatment (after 6 sessions), post-treatment (approximately 14 weeks)
  Spence Children's Anxiety Scale child-report consisting of 38 items rated from 0 (never) to 3 (always) summed to a total score of 0 (no symptoms) to 108 (most severe).

OTHER OUTCOMES:
Change in functioning per parent | Baseline, mid-treatment (after 6 sessions), post-treatment (approximately 14 weeks)
  Children's Sheehan Disability Scale (parent report) consisting of 5 items rated from 0 (not at all) to 10 (very, very much) summed to total score ranging from 0 (no interference) to 50 (severe interference).
Change in functioning per child | Baseline, mid-treatment (after 6 sessions), post-treatment (approximately 14 weeks)
  Children's Sheehan Disability Scale (child report) consisting of 3 items rated from 0 (not at all) to 10 (very, very much) summed to total score ranging from 0 (no interference) to 30 (severe interference).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Whiteside, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Current upon request. Determining how to make data more easily accessible.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following publication of results. Indefinitely by request.
Access Criteria: Approval of analysis plan

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT05777161/Prot_SAP_000.pdf